CLINICAL TRIAL: NCT05699109
Title: Short Versus Long-Acting Erythropoiesis Stimulating Agents for Anemia Management in Egyptian Hemodialysis Patients
Brief Title: Erythropoiesis Stimulating Agents for Anemia Management in Egyptian Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Salma Magdy Abdelfattah, Teaching Assistant, Helwan University
Other Study IDs: Anemia in CKD
Record Dates: First submitted 2023-01-14; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Anemia of Chronic Kidney Disease; Chronic Renal Failure; Chronic Renal Failure Anemia
Keywords: Short / Long-acting ESAs; Hemodialysis; Anemia; Chronic renal failure; Pharmacoeconomics
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aranesp group: Aranesp group: patients received darbepoetin alpha prefilled syringe subcutaneously once weekly or biweekly
- Eprex group: Eprex group: patients received epoetin alpha prefilled syringe subcutaneously one to three times per week

SUMMARY:
This observational study aims to compare long-acting darbepoetin alpha versus short-acting epoetin alpha erythropoietin-stimulating agents in Egyptian hemodialysis patients. The main questions aim to answer are:

* What are the effectiveness and safety of long- acting versus short-acting erythropoietin-stimulating agents in Egyptian hemodialysis patients?
* What is the cost-effectiveness of long- acting versus short-acting erythropoietin-stimulating agents in Egyptian hemodialysis patients?

Participants will be divided into 2 groups; epoetin alfa (short-acting ESA), Eprex group, and darbepoetin alfa (long-acting ESA), Aranesp group for six month study period.

DETAILED DESCRIPTION:
Anemia, the most prevalent and dangerous complication of chronic kidney disease, is caused when the kidney is unable to produce enough erythropoietin to promote the creation of red blood cells (CKD). Anemia from CKD is linked to higher mortality, cardiovascular disease, exhaustion, dyspnea, and a lower quality of life for patients.

It has been demonstrated that using erythropoietin-stimulating drugs (ESAs) in treating renal anemia increases survival, lowers cardiovascular morbidity, and improves the quality of life.

Epoetin alfa (EPO), an ESA with a shorter half-life, and darbepoetin alfa (DPO), are the two ESAs used in hemodialysis centers the most frequently in Egypt (longer half life ) Epoetin alfa is dosed one to three times per week, whereas darbepoetin alfa is dosed once per week or every two weeks.

Compared to epoetins, darbepoetin alfa's extended dose interval may benefit patients and their medical professionals.

Despite the fact that ESAs save CKD patients from needing blood transfusions, clinical trials, meta-analyses, and mortality hazards with ESAs targeting high hemoglobin levels have been shown. A higher ESA dose may be linked to cardiovascular problems and all-cause mortality independent of hemoglobin level.

Darbepoetin alfa has a lower risk of side effects because it only requires 35% of the dosage of epoetin alfa to attain the same target hemoglobin level. Darbepoetin alfa also has an advantage over epoetin alfa in that it makes it easier for the body to mobilize iron into the bone marrow to cause successful erythropoiesis, which may shield the body from any potential negative effects from having too much iron stored there. Despite this, the medication that Egyptian hemodialysis centers use the most is (EPO). This study compares (DPO) and (EPO) to determine which should be utilized based on efficacy, safety, and cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been stable and undergoing hemodialysis three times per week for at least three months
* Age must be 18 or older
* Patients who had been receiving a single form of ESA treatment for at least three months before the study's launch.

Exclusion Criteria:

* altered the type of ESA therapy; 2) underwent significant surgery; or (3) received RBC transfusions
* failed to adhere to dialysis therapy, as shown by missing more than two appointments each month.
* have COVID-19 infection.
* had cancer.
* underwent a kidney transplant
* were pregnant or nursing mothers
* were not followed up for the full six-month research period.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients that followed the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching the target Hemoglobin in each group. | baseline to six months
  Assess the percentage of patients reaching the target Hemoglobin (10-11.5 g/dl) in each group during the study period.

SECONDARY OUTCOMES:
Analyze the cost-effectiveness of long-acting (DPO) versus short-acting (EPO) erythropoietin-stimulating agents in hemodialysis patients. | baseline to six months
  Determine which of the 2 regimen groups is the cost-saving regimen by the cost-effectiveness analysis to examine both the costs and health outcomes of long-acting (DPO) versus short-acting (EPO) erythropoietin-stimulating agents in hemodialysis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Abdel-Hameed Ibrahim Ebid, Professor, Principal Investigator — Faculty of Pharmacy, Helwan University; Amira Mohamed El-Sawy, Lecturer, Study Director — Faculty of Pharmacy, Helwan University; Hazem Ayoub, Lecturer, Study Director — Faculty of Medicine, Al Azhar University
Locations (1):
- the Memorial Souad Kafafi University Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernieh B, Abouchacra S, Boobes Y, Al Hakim MR, Nagelkerke N, Chaaban A, Ahmed M, Hussain Q, Jack HE, Abayechi F, Khan I, Gebran N. Comparison between short- and long-acting erythropoiesis-stimulating agents in hemodialysis patients: target hemoglobin, variability, and outcome. Int Urol Nephrol. 2014 Feb;46(2):453-9. doi: 10.1007/s11255-013-0640-7. Epub 2014 Jan 22. PMID 24448756
- [Background] Biggar P, Ketteler M, Hennemann H, Domling R. Switch of ESA therapy from darbepoetin-alpha to epoetin-beta in hemodialysis patients: a single-center experience. Clin Nephrol. 2008 Mar;69(3):185-92. doi: 10.5414/cnp69185. PMID 18397717
- [Background] Sinha SD, Bandi VK, Bheemareddy BR, Thakur P, Chary S, Mehta K, Pinnamareddy VR, Pandey R, Sreepada S, Durugkar S. Efficacy, tolerability and safety of darbepoetin alfa injection for the treatment of anemia associated with chronic kidney disease (CKD) undergoing dialysis: a randomized, phase-III trial. BMC Nephrol. 2019 Mar 13;20(1):90. doi: 10.1186/s12882-019-1209-1. PMID 30866856
- [Background] Chen N, Xing C, Niu J, Liu B, Fu J, Zhao J, Ni Z, Wang M, Liu W, Zhao J, Zhong L, Wu X, Li W, Chen Y, Shi W, Chen J, Yin A, Fu P, Wang R, Jiang G, Hou F, Ding G, Chen J, Xu G, Kondo Y, Su Y, Mei C. Darbepoetin alfa injection versus epoetin alfa injection for treating anemia of Chinese hemodialysis patients with chronic kidney failure: A randomized, open-label, parallel-group, non-inferiority Phase III trail. Chronic Dis Transl Med. 2022 Mar 29;8(1):59-70. doi: 10.1002/cdt3.13. eCollection 2022 Mar. PMID 35620165
- [Derived] Soliman AE, Magdy S, Ayoub HS, Ebid AI. Short versus long-acting erythropoiesis-stimulating agents for anemia management in Egyptian hemodialysis patients. Qatar Med J. 2024 Mar 11;2024(1):16. doi: 10.5339/qmj.2024.16. eCollection 2024. PMID 38567102